CLINICAL TRIAL: NCT02065206
Title: Spreading Teen-Recorded Inspirational Videos to Engage Schoolmates
Acronym: STRIVES
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-0848; 1R01GM107721-01 (NIH)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Communication
Keywords: Focus groups; Underrepresented Minorities; Social Media; Clinical Research Careers
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
While few students may consider a career in research at baseline, receiving information from peers via online social networks represents a potential way of reaching underserved minority students.

This study addresses a critical problem in the process to diversify the pipeline of clinical researchers - how to cultivate baseline interest in research among high achieving youth before they participate in pipeline programs. We will seek to challenge existing paradigms of studying effectiveness of interventions to promote entry of minority youth into clinical research careers through testing a novel social media campaign that aims to increase interest in research careers among schoolmates of students in a pipeline program. We are testing the use of of peer-created and inspired videos about career choice as a novel way to develop messages that have potential to influence teens.

Should this research program be successful, it will yield valuable insights for researchers and educators who are attempting to train minority students about the importance of involving youth in creating materials to recruit and retain minorities into pipeline programs and educational programs targeted towards clinical research.

DETAILED DESCRIPTION:
Despite several decades of effort that have produced meaningful insights into factors affecting the entry of minority students into careers in health research, there is still a great need to further promote entry of minority students into health research. Research we have done building on broader research on how minority youth select careers has shown that when minority students are interested in career in health research, a dedicated program with realistic career experiences and multi-tiered mentors can increase knowledge, attitudes and behaviors needed for a career in health research. However, we found that such programs are much less effective if students do not enter them with a pre-existing interest in careers in health research. Unfortunately, very little is known about how to increase the interest in careers in health research. Research is badly needed on interventions that can "prime the pump" for pipeline programs by increasing the number of minority students with interest in careers in health research.

Studies from adolescent health education suggest that messages that have the potential to change people's attitudes and behaviors often originate from a trusted peer. A peer messenger is often more easily able to relate to an individual and understand the unique pressures that an individual may face in changing their behavior. This is especially true in teens, who are more likely to value the opinion of and seek to emulate their peers compared to adults. While peer pressure is often cast as a negative phenomenon among teens, the use of positive modes of peer pressure to change behavior among teens is gaining in popularity. For example, positive peer pressure has been used in many youth-to-youth messaging campaigns related to difficult to change behaviors such as alcohol and drug abuse or safe sex.

Peer online social networks may be a potential way to increase interest in careers in health research among underrepresented minority students. The explosion of social media and smartphones has facilitated the creation of social networks online, a well-documented way for teenagers to interact with each other and to obtain information. According to the Pew Internet Project, nearly three quarters of online teens and an equal number of young adults use social network sites. Moreover, roughly 85% of teens who use social networks are active participants in the site, and engage in activities such as posting comments on a friend's profile page, or underneath a friend's picture. Nearly 40% of teens report sharing content online that they created personally. The use of self-created videos has exploded with the creation of popular media-sharing websites, such as YouTube and roughly one third of teens report sharing videos.

Interestingly, there is reason to believe that online social networking interventions that aim to boost career interests would be more effective for underrepresented racial and ethnic groups as well as teens from low income families than for whites. First, data suggests that online social network use is higher among teens from low-income families (those earning less than $30,000 annually) than in teens from wealthier households (80% vs. 70%). Moreover, minority families are more likely to access the internet remotely through mobile devices such as cell phones than whites. Together, this data highlights the enormous potential for online social media interventions to influence career interest and engagement in minority youth.

One promising solution to increase interest in clinical research careers among high achieving youth at a time when career decision making is easily influenced is through the spreading video messages crafted by youth for youth through social media. Therefore, the specific aims of this proposal are the following:

Specific Aim 1: To engage high achieving minority youth enrolled in an intensive pipeline clinical research program in performing focus groups and surveys of their peers to characterize what types of messages would be most likely to motivate their peers to consider a career in clinical research

Specific Aim 2: To engage high-achieving minority youth participating in a pipeline clinical research program in a social media campaign in which they will create a short video to promote interest in clinical research careers and spread it to their schoolmates

Specific Aim 3: To evaluate the reach of social media campaign led by students in a pipeline clinical research program to spread a video they create to improve interest in clinical research careers

Specific Aim 4: To evaluate the effects of a student-led social media campaign on interest in a clinical research career among the schoolmates of students in a pipeline clinical research program

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, the subjects must be between the ages of 15-17 years old. The focus group participants will be recruited from the Collegiate Scholars Program which is a pipeline program for Chicago Public School students.
* The feedback group will be recruited by friends involved in the Teach Research study. They must be named by one of their friends participating in Teach Research.

Exclusion Criteria:

- Participants 18 years or older as well as wards of the state will be excluded from the study.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All subjects enrolled will be under 18 years of age. Subjects 18 and over will not be enrolled. The subjects for this study include two populations of students age 15-17: (1) Collegiate Scholars members to participate in focus groups and (2) feedback group recruited by students involved in TEACH research to view the social media campaign.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Measuring Interest in Clinical Research Careers Among Feedback Group Participants | Every year for four years

SECONDARY OUTCOMES:
Focus Groups | Every year for four years
  Characterize what type of messages would be most likely to motivate peers to consider a career in clinical research.

CONTACTS AND LOCATIONS:
Overall Officials: Vineet M Arora, MD, MAPP, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States